CLINICAL TRIAL: NCT01115218
Title: The Influence of Anterior Chamber Fluid Mediators on the Success Rate of Trabeculectomy
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Arno Hueber, Arno Hueber, University of Cologne
Other Study IDs: MeVeTra-2009
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Glaucoma; Trabeculectomy; Wound Healing
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glaucoma patients
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Procedure: Trabeculectomy — Trabeculectomy with mitomycin C

SUMMARY:
The aim of the study is to investigate whether it is possible to predict the success of trabeculectomy in patients with glaucoma through the examination of mediators of wound healing in anterior chamber fluid. The success rate of trabeculectomy with mitomycin C in the literature is about 75%. This leads on the question why 25% of the patients received trabeculectomy are not sufficient treated and have not a long-term IOP reduction. Precisely this question is to be examined by the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with glaucoma with a trabeculectomy required
* 60 eyes of 60 patients, The ratio of female / male is not involved.
* Eye pressure under local therapy: 20mmHg and above (corrected with pachymetry table).
* age of at least 18 years

Exclusion Criteria:

* all patients not included in the group of inclusion criteria.
* less than 50yl anterior chamber fluid could be collected during the operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the University Eye Hospital of Cologne
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, University of Cologne, Cologne, North Rhine-Westphalia, Germany